CLINICAL TRIAL: NCT00330070
Title: An 8 Week, Randomized, Double-Blind, Parallel Group, Multicenter Trial Comparing the Efficacy and Safety of Oral IPL512,602 to Placebo in Subjects With Moderate to Severe Persistent Asthma Inadequately Controlled on Inhaled Corticosteroids
Brief Title: Control of Asthma Patients Symptomatic on Inhaled Corticosteroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflazyme Pharmaceuticals Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPL512,602-2002; CAPSICS; EudraCT 2006-000840-22
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2007-02-16 (Estimated); Status verified 2007-02

CONDITIONS: Asthma
Keywords: 8-week treatment; oral tablets; persistent moderate to severe asthma; AQLQ; asthma control; quality of life
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: IPL512,602 20 mg once daily
Drug: IPL512,602 Matching Placebo once daily

SUMMARY:
The purpose of the study is to determine whether IPL512,602 is safe and effective for the treatment of asthma symptoms in patients who remain symptomatic on a background therapy of inhaled corticosteroids.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled, parallel group study will include subjects with persistent moderate to severe asthma who require inhaled corticosteroids and inhaled short-acting β2-agonists (SABAs). Subjects who pass screening at Visit 1 will enter a 2-3 week baseline period to confirm stable asthma symptoms and collect baseline data. Subjects will continue with ongoing prescribed treatment during this period, or as modified by the investigator based on clinical judgment. Subjects will use the SABA prescribed for them to alleviate asthma symptoms on an as needed basis throughout the study. If eligible, at Visit 2 subjects will be randomized to treatment with either IPL512,602 (20 mg) daily or placebo in a 1:1 ratio. Randomization in each treatment group will be stratified into two subgroups: those receiving low to medium doses of inhaled corticosteroids (≤500 µg per day fluticasone or equivalent) and those receiving high doses of inhaled corticosteroids (>500 µg per day fluticasone or equivalent). During the 8-week treatment period, subjects will return to the clinic after 1, 2, 4, 6, and 8 weeks of treatment (Visits 3-7). Adverse event data will be collected for 14 days following the last dose administration (Visit 8).

ELIGIBILITY:
Inclusion Criteria:

* a history of persistent asthma for at least the 4 months prior to entry
* require daily inhaled corticosteroids (220-1000 µg fluticasone equivalent per day) for at least 4 weeks prior to randomization and short-acting beta-2-agonist (SABA)
* FEV1 at randomization (without exposure to a SABA for at least 6 hours) must be between 50% and 80% of predicted normal
* reversibility of FEV1 by at least 12% and at least 250 mL following two to four inhalations of a SABA must be demonstrated prior to randomization
* AQLQ(S) score of 4.5 or less at both the screening (Visit 1) and randomization (Visit 2) visits
* patients must meet at least two out of three of the following criteria:

  * overall score minimum of 2 on Asthma Control Questionnaire (ACQ)
  * require rescue SABA use of 2 or more inhalations per day for symptom relief on at least 4 of 7 days during each week of the baseline period
  * nighttime awakenings due to asthma, an average of at least once a week during the baseline period

Exclusion Criteria:

* history of chronic pulmonary diseases other than asthma, including bronchitis, chronic obstructive pulmonary disease (COPD), emphysema, cystic fibrosis, pulmonary tuberculosis, or bronchiectasis
* other asthma therapies:

  * use of long-acting beta-2-agonists within 5 weeks prior to randomization
  * use of leukotriene modulators, theophylline, or muscarinic antagonists within 4 weeks prior to randomization
  * use of injectable or oral corticosteroids within 2 months prior to screening
* requirement for more than 10 inhalations per day of a short-acting beta-2-agonist more than 3 times per week during the baseline period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2006-05; Study Completion 2007-01

PRIMARY OUTCOMES:
Change in AQLQ(S) overall scores from baseline to 8 weeks post-randomization

SECONDARY OUTCOMES:
Change in AQLQ(S) individual domain scores
Change in asthma control
Change in FEV1
Change in morning and evening PEFR
Change in SABA usage
Change in nighttime awakenings
Total number of asthma worsening events
Change in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(S)

CONTACTS AND LOCATIONS:
Overall Officials: Busse William, MD, Principal Investigator — University of Wisconsin, Madison; Jonathan Corren, MD, Principal Investigator — Allergy Research Foundatin, Inc.; Alan Heller, MD, Principal Investigator — San Jose Clinical Research; Edward Kerwin, MD, Principal Investigator — Clinical Research Institute of South Oregon; Y. Hsu, MD, Principal Investigator — West Coast Clinical Trials; Eli Meltzer, MD, Principal Investigator — Allergy and Asthma Medical Group; S. David Miller, MD, Principal Investigator — Northeast Medical Research Associates; Michael J Noonan, Principal Investigator — Allergy Associates Research Center
Locations (8):
- United States (8):
  - West Coast Clinical Trials, Long Beach, California
  - Allergy Research Foundation, Inc., Los Angeles, California
  - Asthma Medical Group & Resarch, San Diego, California
  - San Jose Clinical Research, San Jose, California
  - Northeast Medical Research Associates, Inc, No. Dartmouth, Massachusetts
  - Clinical Research Institute of South Oregaon, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - University of Wisconsin - Madison, Madison, Wisconsin